CLINICAL TRIAL: NCT06372886
Title: Clinical Outcomes of Preservation Versus Resection of Portal/Superior Mesenteric Vein During Pancreaticoduodenectomy in Pancreatic Cancer Patients Who Respond to Neoadjuvant Treatment
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Young Jang, Professor, Seoul National University Hospital
Other Study IDs: 2402-147-1516
Record Dates: First submitted 2024-04-08; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Head Cancer Patients Who Underwent Surgery After Neoadjuvant Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preservation of portal/superior mesenteric vein
  Interventions: Procedure: portal/superior vein resection
- Resection of portal/superior mesenteric vein
  Interventions: Procedure: portal/superior vein resection

INTERVENTIONS:
Procedure: portal/superior vein resection — portal/superior vein resection

SUMMARY:
1. There is a lack of evidence on the need to perform portal/superior mesenteric vein (PV/SMV) resection routinely in pancreatic ductal adenocarcinoma (PDAC) patients with venous involvement who responded to neoadjuvant treatment (NAT).
2. There is no significant differences in R0 rate, 5-year overall survival and recurrence-free survival between the PV/SMV preservation (PVP) group and PV/SMV resection (PVR) group.
3. PVP group showed significantly better 5-year PV/SMV stenosis free survival than the PVR group.
4. We propose that if dissection is possible and there is a high likelihood of achieving R0 resection after NAT, routine PVR may be unnecessary in PDAC patients with venous involvement.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic head cancer patients who underwent surgery after neoadjuvant treatment between January 2012 and December 2022 at Seoul National University Hospital

Exclusion Criteria:

* Metastatic unresectable and locally advanced pancreatic cancer
* Resectable pancreatic cancer without portal/superior mesenteric vein invasion
* Cancer aggravation after neoadjuvant treatment
* Portal/superior mesenteric vein encasing and narrowing after neoadjuvant treatment
* Patients who underwent palliative surgery
* Non-pancreatic ductal adenocarcinoma patients
* Patients who death within 30 days of surgery
* Loss of follow-up patients
* Patients who underwent resection for suspected main artery and adjacent organ invasion

Max Age: 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study retrospectively included 264 pancreatic head cancer patients who underwent surgery after neoadjuvant treatment between January 2012 and December 2022 at Seoul National University Hospital in Korea. Among 264 patients, we included 113 patients with resectable and borderline resectable pancreatic ductal adenocarcinoma with venous involvement who responded to NAT and underwent curative PD.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
5-year overall survival | assessed up to 60months
  from diagnosis to any cause of death
5-year portal/superior mesenteric vein stenosis free survival | assessed up to 60months
  from surgery to stenosis